CLINICAL TRIAL: NCT05454930
Title: Effect of Commute Traffic on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Joel Daniel Kaufman, Professor, Environmental & Occupational Health Sciences, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00001196; K24ES013195 (NIH); RD-83479601 (Other Grant/Funding Number: US Environmental Protection Agency STAR)
Record Dates: First submitted 2015-07-31; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases
Keywords: air pollution; traffic; vascular function; gasoline exhaust; diesel exhaust
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typical Commute (No Intervention): Participants spend two hours in automobile, on heavily trafficked roadways, without active filtration of air pollutants
- Typical Commute, Filtered Air (Other): Participants spend two hours in automobile, on heavily trafficked roadways, with active filtration of air pollutants
  Interventions: Other: Filtered Air

INTERVENTIONS:
Other: Filtered Air — The vehicle is fitted with a (High-Efficiency Particulate Absorbing, HEPA) filter device incorporating a charcoal filter, as well as an augmented cabin filter
  Arms: Typical Commute, Filtered Air

SUMMARY:
The investigators will assess the vascular effects of riding in a car in heavily trafficked roadways, and whether filtering the car's air reduces those effects.

DETAILED DESCRIPTION:
In this double-blind, crossover trial, randomized to order, recruited participants will be screened and then will accompany the study team on three typical commutes on separate days with sufficient washout (i.e., three weeks) between drives. One day this will occur with an effective filter system in the vehicle and the other two days without effective filtration; ineffective filtration is the most typical actual vehicle condition. Subjects will be unaware of the filtration conditions of the commute on that day. Each subject's experimental sessions will occur at the same time of day and will be separated by at least 21 days. The two sessions (either filtered air or traffic-derived entrained air) will be 120 minutes in duration and will encompass routes on heavily traveled roadways in the Seattle area. Before subjects begin the commute trials, they will go through the consent process and a series of screening tests. The study investigators will assess a series of measures regarding vascular function before and after each drive.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* asthma,
* high blood pressure,
* diabetes,
* high cholesterol,
* other chronic conditions requiring ongoing medical care.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Brachial Artery Diameter from Pre-Drive to Post-Drive | 30 minutes before 120 minute driving session; 30 minutes post driving session
  Ultrasound assessment of brachial artery diameter, in millimeters.
Change in Blood Pressure from Pre-Drive to During-Drive and Post-drive | 10 minutes before driving session; 15, 30, 45, 60, 75, 90, 100, 120 minutes following start of (120 minute) driving session; 10 minutes, 1.5 hours, 3.5 hours, 6 hours, 24 hours after end of driving session.
  systolic and diastolic blood pressure measured in mmHg
Change in Retinal Arteriolar Diameter from Pre-Drive to Post-Drive | 30 minutes before 120 minute driving session; 30 minutes post driving session
  measured by retinal photography, image analysis, in micrometers
Gene Expression and DNA methylation | 30 minutes before 120 minute driving session; 30 minutes, 5 hour, and 24 hours post-driving session
  analysis in circulating mononuclear cells; determined via fold change in abundance

SECONDARY OUTCOMES:
circulating stress hormone | 30 minutes before 120 minute driving session; 5 hour and 24 hours post-driving session
  cortisol by chemiluminescence (ng/mL)
complete blood count with differential | 30 minutes before 120 minute driving session; 5 hour and 24 hours post-driving session
  laboratory values for hematologic indices (cells/uL)
inflammatory marker interleukin-6 | 30 minutes before 120 minute driving session; 5 hour and 24 hours post-driving session
  interleukin-6 determined by chemiluminescence (pg/mL)
inflammatory marker c-reactive protein | 30 minutes before 120 minute driving session; 5 hour and 24 hours post-driving session
  C-reactive protein by immunoturbidimetry (ug/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Kaufman, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Young MT, Jansen K, Cosselman KE, Gould TR, Stewart JA, Larson T, Sack C, Vedal S, Szpiro AA, Kaufman JD. Blood Pressure Effect of Traffic-Related Air Pollution : A Crossover Trial of In-Vehicle Filtration. Ann Intern Med. 2023 Dec;176(12):1586-1594. doi: 10.7326/M23-1309. Epub 2023 Nov 28. PMID 38011704